CLINICAL TRIAL: NCT06106425
Title: Diagnostic and Prognostic Criteria of EEG in Neonatal Convulsions at Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eslam Mahrous Mohammedein, Doctor, Assiut University
Other Study IDs: EEG in neonatal convulsions
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: EEC
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EEG — diagnostic tool

SUMMARY:
Diagnostic and prognostic criteria of EEG in neonatal convulsions at Assiut University Children Hospital

DETAILED DESCRIPTION:
The electroencephalogram (EEG) was invented almost 100 years ago and is still a method of choice for many research questions. It is a graphic representation of the difference in voltage between two different cerebral locations plotted over time. The scalp EEG signal generated by cerebral neurons is modified by electrical conductive properties of the tissues between the electrical source and the recording electrode on the scalp, conductive properties of the electrode itself, as well as the orientation of the cortical generator to the recording electrode, (Olejniczak, P et al 2006).

EEG is best used to study the response of the brain to events in the environment or to internal changes during a seizure. EEG is one of the main tools for obtaining electrophysiological information about cerebral function, (Fowle AJ, Binnie CD et al 2000).

Research using neonatal electroencephalography (EEG) has been limited by a lack of a standardized classification system and interpretation terminology.

Electroencephalography (EEG) is an important tool to assess brain function in neonates, for whom clinical observation alone is often insufficient to accurately evaluate cerebral function. EEG is used to assess the severity of brain dysfunction in neonates with known or suspected brain injury; abnormal EEG background features may serve as indicators of unfavorable long-term prognosis, (Wusthoff CJ, Sullivan J et al 2017).

Seizures are the most frequent neurological event in newborns and clinical data suggest that etiology is the dominant factor in long term outcome. However, there are consistent background EEG abnormalities associated to neonatal seizures that are usually related to unfavorable outcome. For example, the burst - suppression pattern may appear related to many neonatal neurological disorders and is associated with early and refractory neonatal seizures, (Nunes ML, Giraldes MM et al 2005).

Also, a normal EEG in a term newborn with hypoxic ischemic encephalopathy (HIE) is associated with good neurological outcome. (Jose A, Matthai J et al 2013).

The chances of survival of preterm infants have increased markedly during recent decades. However, despite this improved survival prognosis, several studies have pointed towards the poor psychomotor outcome of these infants. For example, periventricular leukomalacia is the most common type of hypoxic-ischaemic brain damage causing poor psychomotor development in usually very preterm infants. Diagnostic procedures for detecting brain damage in newborn infants are of two types: bedside and non-bedside techniques. The neuro-developmental outcome is correlated with the number of positive Rolandic sharp waves seen on the EEG recording,

ELIGIBILITY:
Inclusion Criteria:

* - Neonates (< 28 days) presenting with a convulsive attack in the form of a paroxysmal alteration in motor function.

Exclusion Criteria:

* Non- seizure events as Tremors, Jitteriness or Clonus or Neonatal Apnea
* Normal Newborn Behaviour such as stretching, coughing or gagging,
* Physiological Benign Neonatal Myoclonus during sleep

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: 95 cases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
evaluate the role of EEG as a diagnostic as well as prognostic tool in neonatal convulsions. | Baseline
  Diagnostic and prognostic criteria of EEG in neonatal convulsions at Assiut University Children Hospital

REFERENCES:
- [Background] Dereymaeker A, Pillay K, Vervisch J, De Vos M, Van Huffel S, Jansen K, Naulaers G. Review of sleep-EEG in preterm and term neonates. Early Hum Dev. 2017 Oct;113:87-103. doi: 10.1016/j.earlhumdev.2017.07.003. Epub 2017 Jul 12. PMID 28711233